CLINICAL TRIAL: NCT06676852
Title: Feasibility and Acceptability of Primary Palliative Care Intervention in Patients Undergoing Hematopoietic Stem Cell Transplantation
Acronym: Primary PC HCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Society of Transplantation and Cellular Therapy (Unknown)
Responsible Party: Principal Investigator, Richard Andrew Newcomb, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-322
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Hematopoietic Cell Transplant; Hematologic Malignancy
Keywords: palliative care; supportive care; primary palliative care; hematopoietic cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm feasibility clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sentinel, primary palliative care intervention (Experimental): All participants will receive Sentinel, a primary palliative care intervention, in this single-arm feasibility trial. Participants will complete patient-reported assessments at the following time points:
  * Baseline (prior to HCT admission)
  * Week-2 of HCT hospitalization (+/- 3 business days)
  * 1 month post-HCT (+/- 7 business days)
  * 3 months post-HCT (+/- 7 business days)
  Interventions: Behavioral: Primary palliative care

INTERVENTIONS:
Behavioral: Primary palliative care — Enrolled patient participants will receive Sentinel prior to and during their hospitalization for HCT. Prior to HCT, a transplant clinician (nurse practitioner - NP) will conduct a focused PC visit to build rapport, manage expectations regarding HCT, review anticipated symptoms, and discuss illness coping strategies. During the HCT hospitalization, HCT physicians and advanced practice providers will incorporate PC domains into their routine care of patients undergoing HCT.

SUMMARY:
Primary PC - or training HCT clinicians to deliver PC domains as part of routine practice - is an alternative model of supportive care. We have developed Sentinel, a primary PC intervention for HCT clinicians and patients. This study will assess Sentinel's feasibility and acceptability.

DETAILED DESCRIPTION:
Patients hospitalized for hematopoietic cell transplantation (HCT) experience physical and psychological symptoms that lead to a deterioration in quality of life (QOL). Integrating specialty palliative care (PC) reduces physical and psychological symptom burden and improves QOL during HCT hospitalization. However, specialty PC remains unavailable and underused at many HCT centers. Primary PC - or training HCT clinicians to deliver PC domains as part of routine practice - is an alternative model of supportive care. We have developed Sentinel, a primary PC intervention for HCT clinicians and patients. We will train HCT clinicians to deliver PC to patients before and during HCT hospitalization. This study will assess Sentinel's feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Undergoing autologous or allogeneic HCT at MGH

Exclusion Criteria:

* Prior receipt of inpatient specialty palliative care on two prior admissions in the past 6 months.
* Significant uncontrolled psychiatric disorders (psychotic disorder, bipolar disorder, major depression) or other co-morbid disease (dementia, cognitive impairment), which the primary oncologist believes prohibits informed consent or ability to participate in study procedures
* Inability to comprehend English as this is a preliminary/pilot study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Up to Day 90
  We will assess feasibility of Sentinel based on the proportion of eligible patients who enroll and the proportion of enrolled patients retained. Sentinel will be deemed feasible if at least 60% of eligible patients are enrolled in the study and patient retention through study procedures is at least 80%, commonly utilized metrics in PC trials

SECONDARY OUTCOMES:
Acceptability | At Day 30
  The intervention will be acceptable for patients if at least 80% of patients report intervention satisfaction (Client Satisfaction Questionnaire mean greater than or equal 3.0/4.0)

OTHER OUTCOMES:
Quality of Life | Up to Day 90
  We will assess longitudinal quality of life using the Functional Assessment of Cancer Therapy - Bone Marrow Transplantation (FACT-BMT)
Physical Symptoms | Up to Day 90
  We will assess longitudinal physical symptom burden using the Edmonton Symptom Assessment System - Revised (ESAS-r)
Anxiety Symptoms | Up to Day 90
  We will assess longitudinal symptoms of depression with the Hospital Anxiety and Depression Scale (HADS)
Depression Symptoms | Up to Day 90
  We will assess symptoms of depression with the Hospital Anxiety and Depression Scale (HADS)
Post-traumatic stress symptoms | Up to Day 90
  We will assess longitudinal symptoms of post-traumatic stress using the Post-traumatic Stress Checklist-Civilian Version (PCL-C)
Coping | Up to Day 90
  We will use select subscales of the Brief-COPE, a 28-item questionnaire that assess patients' use of 14 methods of coping per a 4-point Likert scale. Coping will be classified as 'Approach-oriented' and 'Avoidant'

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber/Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor, Investigator, or designee. The protocol and statistical analysis plan will be made available on ClinicalTrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the study investigator at richard.newcomb@mgh.harvard.edu